CLINICAL TRIAL: NCT05879471
Title: 68Ga-NY104 PET/CT and 18F-FDG PET/CT in Patients With Metastatic Clear Cell Renal Cell Carcinoma: a Prospective, Single Center, Single Arm, Comparative Imaging Trial
Brief Title: 68Ga-NY104 PET/CT in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCRM
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: 68Ga-NY104; PET/CT; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NY104 PET/CT (Experimental): Each patient will receive one dose of 68Ga-NY104 by intravenous route. Dedicated whole-body PET/CT imaging will be performed.
  Interventions: Diagnostic Test: 68Ga-NY104 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NY104 PET/CT — Participants will be administered a single, intravenous bolus of 68Ga-NY104 The recommended administered activity of 68Ga-NY104 is 1.8-2.2 MBq per kilogram bodyweight, subject to variation that may be required owing to variable elution efficiencies obtained during the lifetime of the 68Ga / 68Ga generator The CT and PET imaging session will begin approximately 45 to 75 minutes after 68Ga-NY104 administration.
  Other Names: 68Ga-NYM005 PET/CT

SUMMARY:
This is a prospective, single-center, single-arm, comparative phase 2 study in patients with metastatic clear cell renal cell carcinoma. The goal is to determine the sensitivity of 68Ga-NY104 PET/CT in patients with metastatic clear cell renal cell carcinoma and compare it with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, comparative phase 2 study in patients with metastatic clear cell renal cell carcinoma. Each patient will receive one dose of 68Ga-NY104 and one dose of 18F-FDG by intravenous route. Dedicated whole-body PET/CT imaging will be performed. PET/CT studies will be interpreted by two readers, both of whom will provide independent, blinded interpretations. Imaging interpretations and a composite reference standard will be used to estimate the sensitivity of each modality. The tumor uptake will also be compared for matched lesions.

39 patients will be recruited in Peking Union Medical College Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Histopathological diagnosis of clear cell renal cell carcinoma
3. Metastatic disease confirmed by histopathology or typical appearance of multifocal metastatic disease
4. Expected survival of at least 6 months
5. ECOG ≤ 2
6. Written informed consent provided for participation in the trial
7. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. On VEGF TKI treatment less than 1 week before 68Ga-NY104 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NY104. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NY104 PET/CT is required.
2. Patients on HIF antagonist treatment < 3 months before 68Ga-NY104 PET/CT. CA9, which encodes carbonic anhydrase IX (CAIX), is one of the genes most strongly upregulated by HIF-1. HIF antagonist, such as Belzutifan, might affect the expression of CAIX and thus the binding of 68Ga-NY104 to tumor. Withdraw of at least 3 months is required for HIF antagonist.
3. Pregnancy or breastfeeding.
4. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Positivity of lesions detected by 68Ga-NY104 PET | From study completion to 1 month after completion
  Any focal accumulation that cannot be explained by physiologic uptake of the 68Ga-NY104 will be interpreted as focal lesion.
Positivity of lesions detected by 18F-FDG PET | From study completion to 1 month after completion
  Any focal accumulation that cannot be explained by physiologic uptake of 18F-FDG will be interpreted as focal lesion.

SECONDARY OUTCOMES:
SUVmax of lesions detected by 68Ga-NY104 PET | From study completion to 1 month after completion
  The tracer uptake in focal lesions is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimentional region of interest (ROI) over the lesion using a threshold of 40% SUVmax.
SUVmax of lesions detected by 18F-FDG PET | From study completion to 1 month after completion
  The tracer uptake in focal lesions is quantified using maximal standard uptake value (SUVmax) by drawing a 3-dimentional region of interest (ROI) over the lesion using a threshold of 40% SUVmax.

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Within 2 years after the publication of the main results
Access Criteria: No limit.